CLINICAL TRIAL: NCT07071805
Title: Prevalence of Varicose Veins Among Petrol Pump Workers
Brief Title: Varicose Veins in Petrol Pump Workers
Status: Completed | Type: Observational
Sponsor: Elite College of Management Sciences, Gujranwala, Pakistan (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-GCUF-079334
Record Dates: First submitted 2025-07-06; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Varicose Veins of Lower Limb
Keywords: Tortous; varicose veins; petrol pump workers
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To check the prevalence of varicose veins among petrol pump workers

DETAILED DESCRIPTION:
A cross-sectional study will be conducted among 323 petrol pump workers, with age 25 to 40 years men which working in different petrol pump stations. Convenience sampling technique will be used for data collection. Data will be collected through Aberdeen Varicose vein Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 25-50 years
* Working for at least 7 hours per day
* Workers who are willing to participate

Exclusion Criteria:

* Arterial diseases of lower limb
* Drug reactions in lower limb
* History of trauma of lower extremity
* Amputated lower limb
* Spinal fractures

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The main objective of the study is to determine the prevalence of varicose veins among petrol pump workers at a specific point in time.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Aberdeen Varicose Vein Questionnaire | 12 weeks
  The Aberdeen Varicose Vein Questionnaire was developed in 2013.This questionnaire is scored from zero to 100, where zero represents a patient with no evidence of varicose veins and 100 represents the most severe problems associated with varicose veins.

CONTACTS AND LOCATIONS:
Overall Officials: Rimza Safdar, DPT, Principal Investigator — Elite College of Management sciences
Locations (1):
- Petrol Pumps, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Naik, C., & Monteiro, P. J. (2024). Prevalence of Varicose Veins among Nurses in a Tertiary Care Hospital: A Descriptive Study. Journal of Health and Allied Sciences NU. — https://www.thieme-connect.com/products/ejournals/html/10.1055/s-0044-1791709
- See also: Salawati, E. M., Alghamdi, N. M., Eissa, G. A., & Almaghrabi, S. J. (2024). Prevalence and Awareness of Varicose Veins in Saudi Arabia, A Cross-Sectional Study. Bahrain Medical Bulletin, 46(2). — https://scholar.google.com/scholar?start=80&q=prevalence+of+varicose+veins+&hl=en&as_sdt=0,5#d=gs_qabs&t=1742106114563&u=%23p%3DSH2Q2mXdAHYJ
- See also: Almutiri, B. M., Alshammari, A. M., Alharbi, S. B., Alsuhaibani, A. N., Alenazi, R. S., Alfarhan, G. K., AlMutairi Sr, B., Alamri, L., Alsuhaibani, A., & Alenazi, R. (2024). Evaluating the prevalence and risk factors of varicose veins in surgeons and ope — https://scholar.google.com/scholar?q=related:olHbZByRu9oJ:scholar.google.com/&scioq=varicose+veins+prevalence+and+Associated+Risk+Factors+among+Women+of+Childbearing+Age+Attending+&hl=en&as_sdt=0,5#d=gs_qabs&t=1741221687085&u=%23p%3DGlL_9S9ZsZcJ